CLINICAL TRIAL: NCT03349801
Title: Development of Novel Clinical Endpoints for Interventional Clinical Trials With a Regulatory and Patient Access Intention in Patients With Intermediate Age-related Macular Degeneration (AMD)
Brief Title: Development of Novel Clinical Endpoints in Intermediate AMD
Acronym: MACUSTAR
Status: Active, not recruiting | Type: Observational
Sponsor: Frank G. Holz (Other)
Collaborators: Bayer (Industry); Moorfields Eye Hospital NHS Foundation Trust (Other); Novartis Pharmaceuticals (Industry); Association for Innovation and Biomedical Research on Light and Image (Other); City, University of London (Other); European Clinical Research Infrastructure Network (Other); La Fondation Voir et Entendre (Unknown); Hoffmann-La Roche (Industry); Radboud University Medical Center (Other); University of Sheffield (Other); University College, London (Other); Carl Zeiss Meditec AG (Industry); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor-Investigator, Frank G. Holz, Prof. Dr. med., University Hospital, Bonn
Organization: University Hospital, Bonn (Other)
Other Study IDs: ECR-AMD-2017-13; MACUSTAR (Other Grant/Funding Number: Innovative Medicines Innitiative)
Record Dates: First submitted 2017-11-10; First posted 2017-11-22 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Age Related Macular Degeneration (AMD)
Keywords: iAMD; biomarker; clinical endpoint
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected in the study for two purposes: biobanking and genetic analysis. Detailed instructions on processing and storage of blood samples are provided in a specific manual that will be provided to the clinical sites. Blood samples are stored in a pseudonimysed form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- no AMD: No interventions
  Interventions: Other: No intervention
- early AMD: No interventions.
  Interventions: Other: No intervention
- intermediate AMD: No interventions.
  Interventions: Other: No intervention
- late AMD: No interventions.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — According to clinical practice.

SUMMARY:
Development of novel clinical endpoints for interventional clinical trials with a regulatory and patient access intention in patients with intermediate age-related macular degeneration (AMD) - MACUSTAR

DETAILED DESCRIPTION:
The purpose of the MACUSTAR clinical study is to develop novel clinical endpoints for clinical trials with a regulatory and patient access intention in patients with intermediate age-related macular degeneration (iAMD). Additional objectives are to characterize the visual impairment in iAMD and its progression, as well as identify risk factors for progression to late stage AMD.

Moreover, MACUSTAR aims to optimize and standardize most relevant existing and/or rapidly available clinical endpoints in:

* visual functional outcomes measures
* structural outcomes measures
* patient reported outcomes measures (PROMs)

The study will be composed by two parts:

* a cross-sectional part to technically evaluate the functional and structural outcome measures to support a biomarker qualification by regulatory authorities and payers; and
* a longitudinal part to assess the prognostic power of changes in retinal sensitivity (as measured by microperimetry) for progression from iAMD to late AMD (nAMD and GA).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion criteria (applicable to all groups)

1. Male and female subjects.
2. Aged 55 - 85 years at baseline.
3. Able and willing to provide written informed consent and to comply with the study protocol visits and assessments.

Intermediate AMD

1. Study eye must have iAMD and,
2. The fellow eye must have iAMD and/or, in addition, extrafoveal GA (no atrophy within the central ETDRS subfield), maximum total GA size is 1.25 mm2.
3. ETDRS letter chart BCVA in the study eye not worse than 72 letters (approximately 20/40 Snellen VA equivalent).
4. All general inclusion criteria.

Late AMD

1. Subjects with bilateral GA, bilateral nAMD or nAMD in one eye and GA in the other.
2. BCVA between 20/80 and 20/200 in study eye.
3. All general inclusion criteria.

Early AMD

1. Subjects with medium drusen > 63μm and ≤ 125μm and no AMD pigmentary abnormalities in both eyes and not signs of intermediate or late AMD.
2. All general inclusion criteria.

No AMD

1. No signs of early, intermediate or late AMD in both eyes.
2. All general inclusion criteria only.

Exclusion Criteria:

General Exclusion criteria (applicable to all groups)

1. Media opacity or eye movement disorder (nystagmus) that interferes with retinal imaging data quality in the opinion of the investigator.
2. Severe ptosis, extraocular motility restriction or head tremor preventing adequate fundus visualization in the opinion of the investigator.
3. Any signs of nAMD or GA (does not apply to the late AMD group).
4. Any concurrent intraocular condition in the study eye (e. g. glaucoma or cataract) that, in the opinion of the investigator would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results.
5. Severe non-proliferative diabetic retinopathy, or proliferative diabetic retinopathy.
6. Any diabetic macular edema or macular disease
7. Ocular disorders in the study eye (i. e., pre-retinal membrane) at the time of enrolment that may confound interpretation of study results and compromise visual acuity.
8. Diagnosis of uncontrolled glaucoma with intraocular pressure of >30 mmHg (despite current pharmacological or non-pharmacological treatment).
9. Known systemic illness which in the opinion of the investigator will prevent from actively participating in the study.
10. Concomitant treatment for AMD in either eye (concomitant use of vitamins/supplements is not excluded; does not apply to the late AMD group).
11. Any periocular or intravitreal injections (IVT) in either eye (does not apply to the late AMD group).
12. Participation in any other interventional trial.
13. Obvious retinal changes due to causes other than AMD (e.g. evidenced by an existing diagnosis of monogenetic macular dystrophies, Stargardt disease, cone rod dystrophy, or toxic maculopathies).
14. Any history of allergies to fluorescein.

Intermediate AMD

1. Any GA in the study eye
2. Any extrafoveal GA larger than 1.25 mm2 in the fellow eye.
3. All general exclusion criteria.

Late AMD

1. All general exclusion criteria only.

Early AMD

1. Intermediate or late AMD (following Beckman classification) in any eye.
2. All general exclusion criteria.

No AMD

1. Early to late AMD (following Beckman classification) in any eye.
2. All general exclusion criteria.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include subjects with no AMD or normal aging changes and subjects with AMD classified in accordance with the international Beckman Classification.
  A total of 750 subjects will be recruited:
  * 300 subjects will participate in the Cross-sectional part:
    * 50 with normal aging changes, no AMD
    * 50 with early AMD,
    * 50 with late AMD
    * 150 with iAMD
  * 650 subjects will participate in the longitudinal part:
    * 600 iAMD
    * 50 early AMD
Sampling Method: Non-Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in best corrected visual acuity (BCVA) using an early treatment diabetic retinopathy study (ETDRS) chart | 3 years from baseline
  standard parameter, tested for comparison (reference variable)
Mean change from baseline in scotopic and mesopic microperimetry sensitivity | 3 years from baseline
Mean change from baseline in low luminance visual acuity (LLVA) | 3 years from baseline
Mean change from baseline in vanishing optotypes visual acuity (VA) | 3 years from baseline
Mean change from baseline in low luminance deficit (LLD) | 3 years from baseline
  LLD = BCVA-LLVA
Mean change from baseline in absolute rod threshold of the dark adaptation test | 3 years from baseline
Mean change from baseline in rod intercept time of the dark adaptation test | 3 years from baseline
Proportion of subjects with progression in dark adaptation deficit beyond coefficient of repeatability structural | 3 years from baseline
Mean change from baseline in the cube root of drusen volume by spectral-domain optical coherence tomography (SD-OCT) | 3 years from baseline
Mean change from baseline in retinal thickness by spectral-domain optical coherence tomography (SD-OCT) | 3 years from baseline
Focal pigmentary changes captured by colour fundus photography (CFP) | 3 years from baseline
Presence of refractile deposits | 3 years from baseline
Presence of intraretinal cystoid spaces | 3 years from baseline
Presence of localized retinal pigment epithelium (RPE) hypertransmission | 3 years from baseline
Presence of localized disruption of ellipsoid zone | 3 years from baseline
Presence of localized subsidence of the outer plexiform layer and the inner nuclear layer | 3 years from baseline
Presence of hyporeflective wedge-shaped bands | 3 years from baseline
Presence of reticular drusen/subretinal drusenoid deposits and associated local changes as determined by multimodal imaging | 3 years from baseline
Changes in localized fundus autofluorescence signal alterations | 3 years from baseline
Proportion of subjects with reduction in drusen volume | 3 years from baseline
Proportion of subjects with study eye that progressed to geogrphic atrophy (GA) and/or neovascular age-related macular degeneration (nAMD) | 3 years from baseline
Proportion of subjects with conversions to late AMD detected with fluorescein angiography (FA) that could be detected with OCT-A (at equipped sites) | 3 years from baseline
Presence of quiescent choroidal neovascularisation (CNV) as assessed by optical coherence tomography angiography (OCT-A) (at equipped sites) | 3 years from baseline
OCT-A findings (at equipped sites) | 3 years from baseline
Mean change from baseline in patient-reported low luminance visual functioning, as measured by the vision impairment in low luminance (VILL) questionnaire, including the domains of reading & accessing information | 3 years from baseline
Mean change from baseline in patient-reported low luminance visual functioning, as measured by the VILL questionnaire, including the domains of Orientation & mobility (incl. driving) | 3 years from baseline
Mean change from baseline in patient-reported low luminance visual functioning, as measured by the VILL questionnaire, including the domains of safety | 3 years from baseline
Mean change from baseline in patient-reported low luminance visual functioning, as measured by the VILL questionnaire, including the domains of socio-emotional well-being | 3 years from baseline
Change in utility index from baseline as measure by the patient-reported outcome measure (PROM) utility index | 3 years from baseline
Mean change from baseline in patient-reported health status and utility using the EQ-5D-5L questionnaire (EuroQol Group) | 3 years from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frank Holz, Prof. Dr. med., Principal Investigator — University Hospital, Bonn
Locations (20):
- Righospitalet Copenhagen, Copenhagen, Denmark
- France (2):
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre d'Investigation Clinique Centre National d'Ophtalmologie des Quinze-Vingts, Paris
- Germany (7):
  - University Hospital Bonn, Bonn
  - University Hospital Cologne, Cologne
  - Department of Ophthalmology, University of Freiburg, Freiburg im Breisgau
  - University Eye Hospital Munich, Munich
  - St. Franziskus Hospital, Münster
  - Universtiy Hospital Tuebingen, Tübingen
  - University Eye Hospital Ulm, Ulm
- Italy (3):
  - Luigi Sacco Hospital, Milan
  - Ospedale San Raffaele, Milan
  - G.B.Bietti Eye Foundation, Rome
- Netherlands (2):
  - Radboud University Medical Centre, Leiden
  - Radboud University Medical Centre, Nijmegen
- Portugal (2):
  - Centre for Clinical Trials, AIBILI, Coimbra
  - Centro Hospitalar de São João, E.P.E., Porto
- United Kingdom (3):
  - Queen's University Belfast, Belfast
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rowen D, Carlton J, McDool E, Holz FG, Zakaria N, Terheyden JH, Finger RP; MACUSTAR Consortium. Psychometric Performance of a New Condition-Specific Preference-Weighted Measure, Vision Impairment in Low Luminance-Utility Index, and EQ-5D-5L in Patients With Age-Related Macular Degeneration: A MACUSTAR Study Report. Value Health. 2025 Jul;28(7):1082-1090. doi: 10.1016/j.jval.2025.04.2155. Epub 2025 Apr 26. PMID 40294859
- [Derived] Terheyden JH, Dunbar HMP, Schmitz-Valckenberg S, Behning C, Martinho C, Luhmann UFO, Sassmannshausen M, Luning A, Miliu A, Aires ID, Basile PG, Batuca J, Schmid M, Moll KP, Zakaria N, Tufail A, Binns A, Crabb DP, Leal S, Finger RP, Holz FG; MACUSTAR consortium. Validating candidate endpoints for intermediate age-related macular degeneration trials in a multi-centre setting-lessons from the MACUSTAR study. Eye (Lond). 2025 Apr;39(6):1031-1039. doi: 10.1038/s41433-024-03568-2. Epub 2025 Feb 5. PMID 39910281
- [Derived] Rowen D, Carlton J, Terheyden JH, Finger RP, Wickramasekera N, Brazier J; MACUSTAR Consortium. Development and Valuation of a Preference-Weighted Measure in Age-Related Macular Degeneration From the Vision Impairment in Low Luminance Questionnaire: A MACUSTAR Report. Value Health. 2024 May;27(5):642-654. doi: 10.1016/j.jval.2024.02.001. Epub 2024 Feb 17. PMID 38369283
- [Derived] Sassmannshausen M, Behning C, Weinz J, Goerdt L, Terheyden JH, Chang P, Schmid M, Poor SH, Zakaria N, Finger RP, Holz FG, Pfau M, Schmitz-Valckenberg S, Thiele S; MACUSTAR Consortium Members. Characteristics and Spatial Distribution of Structural Features in Age-Related Macular Degeneration: A MACUSTAR Study Report. Ophthalmol Retina. 2023 May;7(5):420-430. doi: 10.1016/j.oret.2022.12.007. Epub 2022 Dec 20. PMID 36563964
- [Derived] Garzone D, Terheyden JH, Morelle O, Wintergerst MWM, Sassmannshausen M, Schmitz-Valckenberg S, Pfau M, Thiele S, Poor S, Leal S, Holz FG, Finger RP; MACUSTAR Consortium. Comparability of automated drusen volume measurements in age-related macular degeneration: a MACUSTAR study report. Sci Rep. 2022 Dec 19;12(1):21911. doi: 10.1038/s41598-022-26223-w. PMID 36535990
- [Derived] Terheyden JH, Pondorfer SG, Behning C, Berger M, Carlton J, Rowen D, Bouchet C, Poor S, Luhmann UFO, Leal S, Holz FG, Butt T, Brazier JE, Finger RP; MACUSTAR consortium. Disease-specific assessment of Vision Impairment in Low Luminance in age-related macular degeneration - a MACUSTAR study report. Br J Ophthalmol. 2023 Aug;107(8):1144-1150. doi: 10.1136/bjophthalmol-2021-320848. Epub 2022 Mar 30. PMID 35354561
- [Derived] Terheyden JH, Behning C, Luning A, Wintergerst L, Basile PG, Tavares D, Melicio BA, Leal S, Weissgerber G, Luhmann UFO, Crabb DP, Tufail A, Hoyng C, Berger M, Schmid M, Silva R, Martinho CV, Cunha-Vaz J, Holz FG, Finger RP; MACUSTAR consortium. Challenges, facilitators and barriers to screening study participants in early disease stages-experience from the MACUSTAR study. BMC Med Res Methodol. 2021 Mar 17;21(1):54. doi: 10.1186/s12874-021-01243-8. PMID 33731014
- [Derived] Terheyden JH, Holz FG, Schmitz-Valckenberg S, Luning A, Schmid M, Rubin GS, Dunbar H, Tufail A, Crabb DP, Binns A, Sanchez CI, Hoyng C, Margaron P, Zakaria N, Durbin M, Luhmann U, Zamiri P, Cunha-Vaz J, Martinho C, Leal S, Finger RP; MACUSTAR consortium. Clinical study protocol for a low-interventional study in intermediate age-related macular degeneration developing novel clinical endpoints for interventional clinical trials with a regulatory and patient access intention-MACUSTAR. Trials. 2020 Jul 18;21(1):659. doi: 10.1186/s13063-020-04595-6. PMID 32682441
- See also: Related Info — http://macustar.eu

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT03349801/SAP_000.pdf